CLINICAL TRIAL: NCT04537910
Title: A Randomized, Placebo-Controlled, Participant- and Investigator-Blind, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of LY3819253 Administered Subcutaneously to Healthy Participants
Brief Title: A Study of LY3819253 (LY-CoV555) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18124; J2X-MC-PYAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — bamlanivimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3819253 (Experimental): Participants received single subcutaneous (SC) doses of 150 milligram (mg), 350 mg or 700 mg LY3819253.
  Interventions: Drug: LY3819253
- Placebo (Placebo Comparator): Participants received a single SC dose of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3819253 — Administered SC.
  Other Names: LY-CoV555; Bamlanivimab
  Arms: LY3819253
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of LY3819253 when it is given by injection just under the skin to healthy participants. Blood tests will be done to check how much LY3819253 is in the bloodstream and how long the body takes to eliminate it. Participation could last up to 16 weeks and may include up to six visits to the study center, with a one-week overnight stay.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history and physical examination
* Are willing to follow study procedures, including having nasal or nasopharyngeal swabs collected
* Have a body mass index (BMI) within the range of greater than or equal to (≥)18.5 to less than (<)35 kilograms per square meter (kg/m²)
* Male participants must agree to adhere to contraception restrictions
* Female participants must be of non-childbearing potential

Exclusion Criteria:

* Have or have had known or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Have a history or presence of cardiovascular (including hypertension), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disorders that, in the opinion of the investigator, are capable of

  * Significantly altering the absorption, metabolism, or elimination of drugs
  * Constituting a risk while taking the investigational product, or
  * Interfering with the interpretation of data
* Have significant allergies to humanized monoclonal antibodies (mAbs)
* Have any of the following that are clinically significant:

  * Multiple or severe drug allergies, or
  * Intolerance to topical corticosteroids, or
  * Severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Have had lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Have had breast cancer within the past 10 years
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of current hepatitis C (that is, test positive for anti-hepatitis C antibody with confirmed presence of hepatitis C virus [HCV] ribonucleic acid [RNA])

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo SC: Participants received a single subcutaneous (SC) dose of Placebo.
- 150 Milligram (mg) LY3819253 SC: Participants received a single SC dose of 150 mg LY3819253.
- 350 mg LY3819253 SC: Participants received a single SC dose of 350 mg LY3819253.
- 700 mg LY3819253 SC: Participants received a single SC dose of 700 mg LY3819253.
Period: Overall Study
Arm/Group | Placebo SC | 150 Milligram (mg) LY3819253 SC | 350 mg LY3819253 SC | 700 mg LY3819253 SC
Started | 6 | 5 | 7 | 7
Received at Least One Dose of Study Drug | 6 | 5 | 7 | 7
Completed | 6 | 5 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo SC: Participants received a single SC dose of Placebo.
- 150 mg LY3819253 SC: Participants received a single SC dose of 150 mg LY3819253.
- Total: Total of all reporting groups
Arm/Group | Placebo SC | 150 mg LY3819253 SC | 350 mg LY3819253 SC | 700 mg LY3819253 SC | Total
Number analyzed (Participants) | 6 | 5 | 7 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 7 | 7 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.8) | 46.0 (16) | 45.6 (9.2) | 41.4 (9.2) | 44.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 9
  Male | 3 | 4 | 4 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4 | 8
  White | 6 | 2 | 6 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3819253
Description: PK: AUC[0-∞] of LY3819253
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 15, 29, 60, 85 post-dose
Population: All randomized participants who received at least one dose of LY3819253 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day per milliliter(μg*day/mL)
Arm/Group | 150 mg LY3819253 SC | 350 mg LY3819253 SC | 700 mg LY3819253 SC
Number analyzed (Participants) | 1 | 3 | 3
micrograms*day per milliliter(μg*day/mL) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 259 μg*day/mL | 918 (15) | 1390 (34)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to 85 days)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo SC | 150 mg LY3819253 SC | 350 mg LY3819253 SC | 700 mg LY3819253 SC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 2/5 | 1/7 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC (N=6) | 150 mg LY3819253 SC (N=5) | 350 mg LY3819253 SC (N=7) | 700 mg LY3819253 SC (N=7)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Lilly or Supplier shall publish, discuss, or release data emanating from a study without the other party's express written permission which shall not be unreasonably withheld. Nothing herein shall limit supplier's right to respond to legal inquiries.

DOCUMENTS (2):
  • Study Protocol (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04537910/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04537910/SAP_001.pdf